CLINICAL TRIAL: NCT04875897
Title: KeepMED-away-Obstructive Sleep Apnea Trial: Efficacy and Safety of keepMED Positive Airway Pressure Device in Patients With Obstructive Sleep Apnea - keePaOSA
Brief Title: Efficacy and Safety of keepMED Positive Airway Pressure Device in Patients With Obstructive Sleep Apnea
Acronym: keePaOSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: keepMED Ltd. (Industry)
Collaborators: CRI-The Clinical Research Institute GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-210423-00
Record Dates: First submitted 2021-04-28; First posted 2021-05-06 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-05

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Each subject serves as his/her own control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment with keepMED PAP device (Experimental): Therapy night is performed with the keepMED PAP during a polysomnography in the sleep lab
  Interventions: Device: keepMED PAP device

INTERVENTIONS:
Device: keepMED PAP device — The keepMED PAP device is an automatic, wearable positive airway pressure device indicated for treatment of obstructive sleep apnea. A therapeutic pressure is delivered to the patient upper airway through a nasal interface. It is similar to other marketed positive airway pressure devices with respect to its fundamental use of positive airway pressure for the treatment of sleep apnea as well as with regard to its functional components and accessories (e.g., a PAP unit, a mask/nasal interface, an air filter, tubing, etc.).

SUMMARY:
A prospective, multi-centre, single-arm, open-label, interventional study with a non-marketed medical device.

The primary study objective is to assess the efficacy of the keepMED PAP device on modification of respiratory characteristics in patients with OSA at one therapy night in a sleep lab.

Secondarily, the safety of the use of the device in this setting is assessed.

DETAILED DESCRIPTION:
The study includes a baseline visit, a habituation night, and a therapy night. Both nights will be undertaken in the sleep lab under identical conditions and will include the keepMED PAP therapy activated in parallel to polysomnography (PSG).

Baseline diagnostic PSG, performed within one month prior to enrollment to the study, will be used to assess the device efficacy.

An interim analysis to re-estimate the sample size will be performed after availability of data of 50% enrolled and treated study patients. The sample size will be re-estimated based on the observed changes of AHI in the interim analysis.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years.

Newly diagnosed OSA with AHI ≥ 15 events/hours.

Indication for OSA PAP therapy in routine clinical care according to applicable medical guidelines within one month prior to study enrolment.

Naïve to PAP therapy, i.e. even no PAP therapy during a PSG night.

Weight > 30kg.

Signed informed consent.

Exclusion Criteria:

Body Mass Index (BMI) of ≤20 kg/m² or ≥ 35 kg/m².

Pathologically low blood pressure (systolic ≤90mm Hg; diastolic ≤60 mm Hg).

Current unstable or serious medical conditions (such as angina pectoris, myocardial infarction, cancer, stroke, dementia, congestive heart failure) which based on the physician's judgment might put the patient at high risk.

Mixed and central apnea index ≥ 5 events/hour in PSG without PAP therapy.

Bullous lung disease.

Tracheostomy.

Pneumothorax.

Pneumocephalus.

Cerebrospinal fluid leak.

Current sinus or middle ear infection.

Persistent blockage of one or both nostrils (including nasal septum deviation and nasal polyps) or any other reason that leads to difficulty of breathing through the nose while awake.

Any nasal, facial or head abnormalities that would not allow adequate placement of the device.

Previous diagnosis of insomnia, narcolepsy or periodic limb movement disorder that in the judgment of the clinician could affect sleep quality assessment.

Chronic respiratory disease (COPD, pulmonary fibrosis or asthma) or FEV/FVC ≤ 60% in history.

History of respiratory failure.

Supplemental oxygen is required.

Uvulopalatopharyngoplasty or other surgical procedure to correct apnea.

Acute respiratory infection.

Subject recovered from Covid-19 but suffers from on-going symptoms or when subject's Covid-19 illness history can affect the study outcome based on the physician's judgment.

Pregnancy.

Medication that may alter sleep architecture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2021-09-14 (Estimated); Primary Completion 2022-01-15 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Changes of Apnea Hypopnea Index (AHI) | A single therapy night compared to baseline (conducted approx 1 month before the therapy night)
  Efficacy by means of changes of the AHI comparing baseline measures in a sleep lab night without keepMED PAP therapy with measures during one therapy night in a sleep lab.

SECONDARY OUTCOMES:
Changes in oxygen desaturation index (ODI) | A single therapy night compared to baseline (conducted approx 1 month before the therapy night)
  Changes in ODI comparing baseline measures in a sleep lab night without keepMED PAP therapy with measures during one therapy night in a sleep lab
Changes in arousal index (sleep quality) | A single therapy night compared to baseline (conducted approx 1 month before the therapy night)
  Changes in arousal index comparing baseline measures in a sleep lab night without keepMED PAP therapy with measures during one therapy night in a sleep lab
Number of adverse events | Throughout the study, an average of 2-7 days per subject
  Safety of the device use by means of adverse events in patients using the keepMED PAP device

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Pépin, Prof, Principal Investigator — CHU Michallon Laboratoire EFCR CS 10217